CLINICAL TRIAL: NCT05532813
Title: Evaluation of the Efficacy and Safety of Metformin in the Myotonic Dystrophy Type 1 (Steinert's Disease). A Phase III, Prospective, Multicentre, Randomized, Double-blind Controlled Study
Brief Title: Evaluation of the Efficacy and Safety of Metformin in the Myotonic Dystrophy Type 1 (Steinert's Disease)
Acronym: METFORMYO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP220832; 2023-507660-39-00 (Registry Identifier: EU trial number)
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Steinert's Disease; Myotonic Dystrophy 1; Metformin
Keywords: Steinert's Disease; Myotonic Dystrophy 1; Metformin; Muscle function
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin arm (Experimental): Patients randomized in Metformin arm will take metformin orally.
  Interventions: Drug: Treatment taken
- Placebo receivers (Placebo Comparator): Patients randomized in placebo arm will take placebo orally in the same procedure as metformin taken.
  Interventions: Drug: Treatment taken

INTERVENTIONS:
Drug: Treatment taken — Treatment (Metformin or placebo) will be administered orally and titrated following the same guideline that metformin in diabetic patient: start with a daily dose of 500 mg twice a day, given during or after meals; then increase to 1000 mg twice a day after a week. If digestive tolerance is good, treatment will be increased to a maximum of 1000 mg three times a day i.e. 3000 mg/day after another week.

SUMMARY:
The study team hypothesize that non-diabetic patients with Myotonic dystrophy type I (DM1) will improve their symptoms, especially their motor deficit which is the main feature of the disease, because of the splicing defect correction by metformin.

The primary objective of the study is to evaluate the efficacy of metformin vs placebo, on the improvement of muscle function in patients with DM1 compared to its placebo.

As the secondary objectives, the study aims:

* To evaluate the safety of metformin on patient with DM1.
* To evaluate the efficacy of metformin vs placebo on:

  1. The hand-grip strength;
  2. The thumb-index pinch strength;
  3. The locomotor function;
  4. The respiratory function;
  5. The cardiac function;
  6. The quality of life;
  7. The daily and social activity.

DETAILED DESCRIPTION:
This is a multicenter, national, comparative study comparing the efficacy and safety of metformin and placebo in patients (1:1 ratio between the 2 groups) with DM1.

Population of study participants: patients with biochemically and/or genetically confirmed DM1 disease already followed in the referral and competence departments, as well as new patients.

All patients will be included by a neuromuscular specialist from French centers participating in the research.

Enrolled patients were randomly assigned (71 patients per group with 1:1 ratio) to either metformin therapy or a placebo, using a centralized randomization procedure.

Metformin or placebo will be administered orally and titrated as recommended in diabetic patients. Initial digestive effects (nausea, vomiting and constipation) of metformin that can be observed in the first days. If digestive tolerance is good, treatment will be increased to a maximum of 1000 mg three times a day i.e. 3000 mg/day after another week. In case of bad digestive tolerance, the dosage should be decrease and the maximum tolerated dosage of metformin should be used. The evaluations of muscle function, walking test, respiratory and cardiac function, quality of life, and tolerance will be assessed at M6 and M12, in the neuromuscular centers. With the estimated effect size, we believe that the inclusion capacities evaluated at 8 to 12 patients per center over one year (18 reference centers involved) will allow to determine a significant difference of MFM score 12 months after inclusion. Dose titration, monitoring of side effects and dose adjustments will be assessed at each visit according to the site endocrinologist advice, if necessary.

Statistical analysis: The difference between the score at 12 months and baseline will be compared between treatment groups using the Student T-test.

Secondary efficacy endpoints evaluating the evolution of symptoms will be analyzed using either a GMM or a GEE for continuous and categorical variables, respectively.

Other quantitative variables will be compared using the Student t-test (or a non-parametric test if the distribution remains skewed following transformation), while categorical variables will be analyzed using either the Chi-squared or the Fisher-exact tests.

All efficacy endpoints will be analysed on an intention-to- treat basis and safety endpoints on a per-protocol basis.

All statistical tests will be performed with a level of significance of 5%. No interim analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* DM1 disease confirmed by genetic analysis
* Men and women between 18 and 70 years of age.
* Preserved walking abilities (stick assistance possible)
* MIRS score 3 or 4
* Women of childbearing potential under efficient contraception during treatment
* Patient able to consent
* All patients who have completed and signed the specific information and informed consent form
* Affiliation to a social security system

Exclusion Criteria:

* Pregnant or breast-feeding women
* Men with an intention to conceive a child during the time of the study
* Contraindications to Metformin (hypersensitivity to metformin or to one of the excipients)
* Respiratory:

  * Patient requiring tracheotomy or
  * Patient requiring non-invasive-ventilation: - more than 12 hours per day; - insufficiently ventilated
* Creatinine clearance inferior to 50 ml/min
* Cardiac:

  * Left ventricular ejection fraction below 35%
  * Conduction system disease on the electrocardiogram with PR interval >200 ms or QRS duration >110 ms without a pacemaker or an implantable defibrillator or cardiac electrophysiological study performed over the past 5 years
  * Third-degree or Second degree type II atrioventricular block without a pacemaker or an implantable defibrillator
  * Sustained ventricular tachycardia
* Acute disease that may lead to tissue hypoxia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of muscle function | at baseline and 12 months
  By MFM (Motor Function Measure) scale. The MFM-32 is a widely used sensitive and reliable quantitative functional motor scale, validated for use in various neuromuscular disorders (Bérard et al. 2005) and presenting the advantage to measure precisely, not only the muscle strength but motor function which is the main concern for DM1 patients.

SECONDARY OUTCOMES:
Safety endpoint | through study completion, an average of 30 month
  Any serious adverse event, especially lactic acidosis.
Change of muscle function between baseline and 6 months | at baseline and 6 months
  By the MFM (Motor Function Measure) scale.
The hand-grip strength | baseline, 6 and 12 months
  The hand-grip strength defined by the scores obtained using a manual dynamometry standardized (MyoGrip)
The thumb-index pinch strength | baseline, 6 and 12 months
  The thumb-index pinch strength defined by the scores obtained using a standardized manual dynamometry (MyoPinch)
The locomotor function | baseline, 6 and 12 months
  The locomotor function defined by the scores obtained using the 6 Minutes Walking Test.
The respiratory function | baseline, 6 and 12 months
  The respiratory function, using pulmonary function tests, defined by the Supine Vital Capacity (VC).
The cardiac function | baseline, 6 and 12 months
  The cardiac function, using transthoracic echocardiography, defined by the left ventricular ejection fraction.
Quality of life assessement | baseline, 6 and 12 months
  The quality of life defined by the scores obtained using the quality of life in genetic neuromuscular disease questionnaire (QoLgNMD).
The difference between DM1-ActivC at baseline visit, the visit at 6 months and final visit | baseline, 6 and 12 months
  The activity defined by the scores obtained using the DM1 activity and participation scale for clinical use (DM1-ActivC).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal LAFORÊT, MD, PhD, Principal Investigator — Neurology Department, Raymond Poincaré Hospital, APHP
Locations (1):
- Neurology Department, Raymond-Poincaré hospital - APHP, Garches, France

REFERENCES:
- [Background] Berard C, Payan C, Hodgkinson I, Fermanian J; MFM Collaborative Study Group. A motor function measure for neuromuscular diseases. Construction and validation study. Neuromuscul Disord. 2005 Jul;15(7):463-70. doi: 10.1016/j.nmd.2005.03.004. PMID 16106528
- [Background] Landfeldt E, Nikolenko N, Jimenez-Moreno C, Cumming S, Monckton DG, Faber CG, Merkies ISJ, Gorman G, Turner C, Lochmuller H. Change over time in ability to perform activities of daily living in myotonic dystrophy type 1. J Neurol. 2020 Nov;267(11):3235-3242. doi: 10.1007/s00415-020-09970-6. Epub 2020 Jun 15. PMID 32542526